CLINICAL TRIAL: NCT01188018
Title: Can Motivational Interviewing be Effective for Smoking Cessation?
Brief Title: Testing Counseling Styles to Motivate Smokers to Quit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Delwyn Catley, Professor of Psychology, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00023726; 1R01CA133068-01A2 (NIH)
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Smoking; Tobacco Use; Nicotine Dependence
Keywords: Smoking; Smoking Cessation; Nicotine Dependence; Tobacco Use Cessation; Health Education; Patient Education
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Use Disorder; Smoking Cessation; Tobacco Use Cessation; Health Education | interventions — Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief Advice (Active Comparator)
  Interventions: Behavioral: Brief Advice (BA)
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing (MI)
- Health Education (Active Comparator)
  Interventions: Behavioral: Health Education (HE)

INTERVENTIONS:
Behavioral: Brief Advice (BA) — Participants in this arm will receive a single session of brief advice. A counselor will briefly discuss the risks associated with smoking.
  Arms: Brief Advice
Behavioral: Motivational Interviewing (MI) — Subjects will receive 4 counseling sessions (over 18 weeks) in which their thoughts about their smoking will be discussed. Two of these counseling sessions will be performed in person (weeks 0 and 12) and the remaining two will be over the phone(weeks 6 and 18).
  Arms: Motivational Interviewing
Behavioral: Health Education (HE) — Subjects will receive 4 counseling sessions (over 18 weeks)in which they will receive educational information about the risks of smoking and the benefits of quitting. Two of these counseling sessions will be performed in person (weeks 0 and 12) and the remaining two will be over the phone (weeks 6 and 18).
  Arms: Health Education

SUMMARY:
The purpose of this study is to determine, among a sample of general adult smokers, the effectiveness of three different counseling interventions for motivating quit attempts among smokers not yet ready to quit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Smoke at least once a day for the past 30 days
* Are willing to participate in all study components
* Sufficient language skills in English for counseling and assessments
* Has a home address
* Has a working phone number

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next 6 months
* Currently using a smoking cessation medication
* Currently participating in smoking cessation program
* Motivated to quit smoking
* Planning to quit smoking in the next 2 weeks
* Lives in a home with someone currently enrolled in the study
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quit Attempt(s) | Any time within 26 weeks

SECONDARY OUTCOMES:
Smoking Cessation | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Delwyn Catley, Ph.D., Principal Investigator — University of Missouri, Kansas City
Locations (1):
- University of Missouri-Kansas City, Kansas City, Missouri, United States

REFERENCES:
- [Background] 2008 PHS Guideline Update Panel, Liaisons, and Staff. Treating tobacco use and dependence: 2008 update U.S. Public Health Service Clinical Practice Guideline executive summary. Respir Care. 2008 Sep;53(9):1217-22. No abstract available. PMID 18807274
- [Background] Soria R, Legido A, Escolano C, Lopez Yeste A, Montoya J. A randomised controlled trial of motivational interviewing for smoking cessation. Br J Gen Pract. 2006 Oct;56(531):768-74. PMID 17007707
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Derived] Grobe JE, Goggin K, Harris KJ, Richter KP, Resnicow K, Catley D. Race moderates the effects of Motivational Interviewing on smoking cessation induction. Patient Educ Couns. 2020 Feb;103(2):350-358. doi: 10.1016/j.pec.2019.08.023. Epub 2019 Aug 18. PMID 31466882
- [Derived] Bani-Yaghoub M, Elhomani A, Catley D. Effectiveness of motivational interviewing, health education and brief advice in a population of smokers who are not ready to quit. BMC Med Res Methodol. 2018 Jun 13;18(1):52. doi: 10.1186/s12874-018-0511-0. PMID 29895280
- [Derived] Harris KJ, Bradley-Ewing A, Goggin K, Richter KP, Patten C, Williams K, Lee HS, Staggs VS, Catley D. Recruiting unmotivated smokers into a smoking induction trial. Health Educ Res. 2016 Jun;31(3):363-74. doi: 10.1093/her/cyw018. Epub 2016 Apr 13. PMID 27081187
- [Derived] Catley D, Goggin K, Harris KJ, Richter KP, Williams K, Patten C, Resnicow K, Ellerbeck EF, Bradley-Ewing A, Lee HS, Moreno JL, Grobe JE. A Randomized Trial of Motivational Interviewing: Cessation Induction Among Smokers With Low Desire to Quit. Am J Prev Med. 2016 May;50(5):573-583. doi: 10.1016/j.amepre.2015.10.013. Epub 2015 Dec 23. PMID 26711164
- [Derived] Catley D, Harris KJ, Goggin K, Richter K, Williams K, Patten C, Resnicow K, Ellerbeck E, Bradley-Ewing A, Malomo D, Liston R. Motivational Interviewing for encouraging quit attempts among unmotivated smokers: study protocol of a randomized, controlled, efficacy trial. BMC Public Health. 2012 Jun 19;12:456. doi: 10.1186/1471-2458-12-456. PMID 22713093
- See also: KC Quest — http://cas.umkc.edu/kcquest